CLINICAL TRIAL: NCT01143532
Title: Role of Donor Genetics and Recipient Genetics in Kidney Transplant Outcomes
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100135; 10-DK-0135
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Kidney Disease; Kidney Transplantation; Kidney Failure, Chronic
Keywords: African-Americans; MYH9; Chronic Allograft Nephropathy; Chronic Kidney Disease; Proteinuria; Natural History; Kidney Disease; Kidney Transplant; African-American
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney transplant donor of black African descent.: Kidney transplant donor of black African descent.
- Kidney transplant recipient of black African descent: Kidney transplant recipient of black African descent.

SUMMARY:
Background:

- Genetic variation in a particular chromosome is a major contributor to the increased risk for kidney disease that is common in people of African descent, although the specific gene, mutations, and other aspects of the variations remain to be determined. By studying the outcomes of kidney transplant in donors and recipients of African descent, researchers hope to better understand the effects of this genetic variation on the success of kidney transplants.

Objectives:

- To examine possible connections between genetic variations and kidney transplant outcomes for donors and recipients.

Eligibility:

* Participants in kidney transplant where both donor and recipient were of black African descent.
* Eligible transplants include both living donor and deceased donor.

Design:

* The study will involve one visit of up to 8 hours.
* All participants will provide a detailed personal and family medical history.
* All participants will provide blood and urine samples, including a 24-hour urine collection, to test kidney function and collect material for genetic testing.
* Donor participants will also have a magnetic resonance imaging (MRI) scan of their remaining kidney.

DETAILED DESCRIPTION:
Genetic variation in the region of MYH9 and APOL1, located on chromosome 22, is a major contributor to the increased risk for kidney disease that characterizes African descent populations, although the specific gene, causative mutations, and the molecular and cellular mechanisms remain to be determined. We propose to study the role of MYH9 and APOL1 genetic variation, as well as other genes, in renal transplant, including the effect of donor genotype on recipient outcomes and on donor outcomes. Additional exploratory studies will address 1) whether variation in other donor genes might contribute to donor and recipient outcomes, which we may address with candidate gene studies or a genome-wide association study and 2) whether recipient genotype contributes to recipient outcomes, which we will address in similar ways.

MULTICENTER STUDY. We will identify 300 kidney transplant dyads (donor/recipient pairs), in which both individuals were of African descent and the kidney transplants were performed between 1995 and 2006. We will include 150 living donor transplants (selected on the basis of the ability to locate the surviving living donor and their willingness to participate) and 150 deceased donor transplants (selected at random, to minimize survival bias of the allograft). All subjects sign consents that are identical or similar to the NIH consent.

RECIPIENT OUTCOMES. We hypothesize that genetic variants in the kidney donor genome and secondarily in recipient genome might contribute to kidney recipient outcomes. We will obtain kidney donor genotypes using blood from surviving living donors or using transplant kidney biopsy DNA from now-deceased living donors, and we will obtain deceased donor genotypes by using transplant kidney biopsies. We will obtain recipient DNA, when available, from surviving recipients or from tissues obtained from deceased recipients. We will carry out Cox proportional hazards analysis to test the primary hypothesis, that donor MYH9 and APOL1 genotype influences allograft survival. We will also develop a multivariable model to predict last follow-up glomerular filtration rate, incorporating factors known to influence transplant outcomes and examining the effect of donor MYH9 and APOL1 genotype. In exploratory studies, we determine whether recipient genetic variants influence recipient outcomes.

DONOR OUTCOMES. We hypothesize that genetic variants in the kidney donor affect kidney donor outcomes. While kidney donors do not have an increased risk of chronic kidney disease compared to the general population, they do have an increased prevalence of microalbuminuria. Furthermore, the extent of compensatory renal hypertrophy appears to differ among individuals. We wish to determine whether MYH9 and APOL1 genotype affects these outcomes, as well as the uncommon occurrence of overt kidney disease after kidney donation. CLINICAL IMPLICATIONS. We believe that that these studies will expand our knowledge of how donor genotypes influence kidney transplant outcomes for both donors and recipients.

COLLABORATIVE STUDY. In separate but related studies, we will work with various collaborators who pursuing similar question under research protocols that they have generated and for which they have local IRB approvals. We will receive from these collaborators materials for preparation of DNA, from which we will genotype APOL1 and other genes known or hypothesized to be related to donor and recipient transplant outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

We will study 300 African American kidney transplant dyads.

INCLUSION CRITERIA FOR DYADS:

1. African descent donor and African descent recipient
2. Kidney transplant performed Jan 1995 - Dec 2006.
3. First kidney transplant
4. Kidney only transplant (excluding transplant of any other organ at any other time).

EXCLUSION CRITERIA:

1. We will exclude donors whose kidneys were used in transplants in which two organs were transplanted, e.g. pancreas and kidney, either simultaneously or at separate times. We will exclude donors whose kidneys were used in second or subsequent transplants. Rationale: dual organ transplants and serial transplants are more complicated clinical situations and renal allograft survival may be shorter and thus not comparable with other kidney transplants.
2. We will exclude recipients who had HIV, hepatitis B or hepatitis C infection diagnosed either before or after the kidney transplant.
3. Children
4. Pregnant women will be excluded but invited to participate after delivery. The rationale is the renal function is altered during pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will identify 300 kidney transplant dyads (donor/recipient pairs), which both individuals were of African descent and the kidney transplants were performed between 1995-2006. We hypothesize that genetic variants in the kidney donor affect kidney donor outcomes. Kidney donors have an increased prevalence of microalbuminuria.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-08-12 (Actual); Primary Completion 2015-10-19 (Actual); Study Completion 2015-10-19 (Actual)

PRIMARY OUTCOMES:
Whether variation in other donor genes might contribute to donor and recipient outcomes | 1995-2006
  Will identify 300 kidney transplant dyads (donor/recipient pairs), which both individuals were of African descent and the kidney transplants were performed between 1995-2006. We hypothesize that genetic variants in the kidney donor affect kidney donor outcomes. Kidney donors have an increased prevalence of microalbuminuria.

SECONDARY OUTCOMES:
Whether recipient genotype contributes to recipient outcomes. | 1995-2006
  We hypothesize that genetic variants in the kidney donor genome and secondarily in recipient genome might contribute to kidney recipient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-DK-0135.html